CLINICAL TRIAL: NCT01531673
Title: A Phase 2, Multicenter, Double-Blinded, Placebo Controlled Study to Evaluate Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of VX-661 Monotherapy and VX-661/Ivacaftor Cotherapy in Subjects With Cystic Fibrosis, Homozygous or Heterozygous for the F508del-CFTR Mutation
Brief Title: Study of VX-661 Alone and in Combination With Ivacaftor in Subjects Homozygous or Heterozygous to the F508del-Cystic Fibrosis Transmembrane Conductance Regulator(CFTR) Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX11-661-101; 2011-003821-93 (EudraCT Number)
Record Dates: First submitted 2012-02-01; First posted 2012-02-13 (Estimated); Results first posted 2018-04-13 (Actual); Last update posted 2018-04-13 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — tezacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (13):
- Group 1-6d Combined: Placebo (Placebo Comparator): All participants in group 1, 2a, 2b, 3a, 3b, 4, 5a, 5b, 6a and 6d who received placebo matched to VX-661 tablet and/or placebo matched to ivacaftor tablet for up to 28 days.
  Interventions: Drug: Placebo matched to VX-661; Drug: Placebo matched to ivacaftor
- Group 1: VX-661 10 mg qd (Experimental): All participants in group 1 who received VX-661 10 milligram (mg) tablet orally once daily (qd) for up to 28 days.
  Interventions: Drug: VX-661
- Group 2a: VX-661 30 mg qd (Experimental): All participants in group 2a who received VX-661 30 mg tablet orally qd and placebo matched to Ivacaftor tablet every 12 hours (q12h) for up to 28 days.
  Interventions: Drug: VX-661; Drug: Placebo matched to ivacaftor
- Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h (Experimental): All participants in group 2b who received VX-661 10 mg tablet qd and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- Group 3a: VX-661 100 mg qd (Experimental): All participants in group 3a who received VX-661 100 mg tablet orally qd and placebo matched to Ivacaftor tablet q12h for up to 28 days.
  Interventions: Drug: VX-661; Drug: Placebo matched to ivacaftor
- Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h (Experimental): All participants in group 3b who received VX-661 30 mg tablet qd and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h (Experimental): All participants in group 4 who received VX-661 100 mg tablet qd and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- Group 5a: VX-661 150 mg qd (Experimental): All participants in group 5a who received VX-661 150 mg tablet orally qd for up to 28 days.
  Interventions: Drug: VX-661
- Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h (Experimental): All participants in group 5b who received VX-661 150 mg tablet qd and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h (Experimental): All participants in group 6a who received VX-661 100 mg tablet qd and Ivacaftor 50 mg tablet q12h orally for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h (Experimental): All participants in group 6d who received VX-661 50 mg tablet and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor
- Group 7: Placebo (Placebo Comparator): All participants in group 7 who received placebo matched to VX-661 tablet orally qd in combination with physician-prescribed Kalydeco (Ivacaftor) for up to 28 days.
  Interventions: Drug: Ivacaftor; Drug: Placebo matched to VX-661
- Group 7: VX-661 100 mg qd (Experimental): All participants in group 7 who received VX-661 100 mg tablet orally qd in combination with physician-prescribed Kalydeco (Ivacaftor) for up to 28 days.
  Interventions: Drug: VX-661; Drug: Ivacaftor

INTERVENTIONS:
Drug: VX-661
  Arms: Group 1: VX-661 10 mg qd; Group 2a: VX-661 30 mg qd; Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h; Group 3a: VX-661 100 mg qd; Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h; Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h; Group 5a: VX-661 150 mg qd; Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h; Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h; Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h; Group 7: VX-661 100 mg qd
Drug: Ivacaftor
  Arms: Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h; Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h; Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h; Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h; Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h; Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h; Group 7: Placebo; Group 7: VX-661 100 mg qd
Drug: Placebo matched to VX-661
  Arms: Group 1-6d Combined: Placebo; Group 7: Placebo
Drug: Placebo matched to ivacaftor
  Arms: Group 1-6d Combined: Placebo; Group 2a: VX-661 30 mg qd; Group 3a: VX-661 100 mg qd

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) effects of VX-661 alone and when coadministered with ivacaftor in participants with cystic fibrosis (CF) who are homozygous or heterozygous for the F508del-CFTR mutation.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, multicenter, double-blinded, placebo-controlled, study of VX-661 monotherapy, and VX-661/ivacaftor co-therapy in participants with CF who are homozygous or heterozygous for the F508del CFTR mutation.

This study is separated into seven groups: Group 1-7, respectively. Approximately 180 participants were randomized in a ratio of 4:1; active drug to matching placebo in each group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with confirmed diagnosis of CF
* Must have the F508del-CFTR gene mutation in both alleles (Groups 1, 2, 3, 4, 5, 6). Group 7 participants must have the F508del-CFTR mutation on 1 allele, and gating mutation G551D on the second allele and have been on their physician prescribed 150 mg KalydecoTM q12h (commercially available ivacaftor) for at least 28 days at the Screening Visit.
* Forced expiratory volume in 1 second(FEV1) 40% to 90% (inclusive) of predicted normal for age, gender, and height (Knudson standards) at screening
* Weight >40 kg and BMI >18.5
* Participants of child-bearing potential and who are sexually active must meet the contraception requirements.

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 4 weeks before Study Day 1.
* History of solid organ or hematological transplantation
* Participation in a clinical study involving administration of either an investigational or a marketed drug within 30 days or 5 terminal half-lives (whichever is longer) before screening
* History of alcohol, medication, or illicit drug abuse within 1 year prior to screening
* Pregnant, breast-feeding, or not willing to follow contraception requirements

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2012-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Donaldson, MD, Principal Investigator — University of North Carolina
Locations (36):
- United States (19):
  - Vertex Investigational Site, Birmingham, Alabama
  - Vertex Investigational Site, Oakland, California
  - Vertex Investigational Site, Boise, Idaho
  - Vertex Investigational Site, Chicago, Illinois
  - Vertex Investigational Site, Boston, Massachusetts
  - Vertex Investigational Site, Grand Rapids, Michigan
  - Vertex Investigational Site, Kansas City, Missouri
  - Vertex Investigational Site, Long Branch, New Jersey
  - Vertex Investigational Site, New Hyde Park, New York
  - Vertex Investigational Site, Chapel Hill, North Carolina
  - Vertex Investigational Site, Cincinnati, Ohio
  - Vertex Investigational Site, Columbus, Ohio
  - Vertex Investigational Site, Oklahoma City, Oklahoma
  - Vertex Investigational Site, Hershey, Pennsylvania
  - Vertex Investigational Site, Pittsburgh, Pennsylvania
  - Vertex Investigational Site, Charleston, South Carolina
  - Vertex Investigational Site, Salt Lake City, Utah
  - Vertex Investigational Site, Burlington, Vermont
  - Vertex Investigational Site, Seattle, Washington
- Canada (4):
  - Vertex Investigational Site, Calgary, Alberta
  - Vertex Investigational Site, Vancouver, British Columbia
  - Vertex Investigational Site, Halifax, Nova Scotia
  - Vertex Investigational Site, Toronto, Ontario
- Germany (8):
  - Vertex Investigational Site, Erlangen, Bavaria
  - Vertex Investigational Site, Frankfurt am Main, Hesse
  - Vertex Investigational Site, Hanover, Lower Saxony
  - Vertex Investigational Site, Cologne, North Rhine-Westphalia
  - Vertex Investigational Site, Berlin
  - Vertex Investigational Site, Bochum
  - Vertex Investigational Site, Jena
  - Vertex Investigational Site, Munich
- United Kingdom (5):
  - Vertex Investigational Site, Cambridge, Cambridgeshire
  - Vertex Investigational Site, London, Greater London
  - Vertex Investigational Site, Manchester, Greater Manchester
  - Vertex Investigational Site, Southhampton, Hampshire
  - Vertex Investigational Site, Cardiff, Vale of Glamorgen

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 194 participants were randomized of which 190 participants were treated.
Groups:
- Group 7: Placebo: All participants in group 7 who received placebo matched to VX-661 tablet orally qd in combination with physician-prescribed Kalydeco for up to 28 days.
- Group 7: VX-661 100 mg qd: All participants in group 7 who received VX-661 100 mg tablet orally qd in combination with physician-prescribed Kalydeco for up to 28 days.
Period: Overall Study
Arm/Group | Group 1-6d Combined: Placebo | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 7: Placebo | Group 7: VX-661 100 mg qd
Started | 33 | 8 | 8 | 18 | 8 | 19 | 17 | 9 | 17 | 19 | 16 | 4 | 14
Completed | 33 | 7 | 8 | 17 | 7 | 18 | 17 | 9 | 17 | 18 | 16 | 4 | 14
Not Completed | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1: VX-661 10 mg qd: All participants in group 1 who received VX-661 10 mg tablet orally qd for up to 28 days.
- Group 2a: VX-661 30 mg qd: All participants in group 2a who received VX-661 30 mg tablet orally qd and placebo matched to Ivacaftor tablet q12h for up to 28 days.
- Total: Total of all reporting groups
Arm/Group | Group 1-6d Combined: Placebo | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 7: Placebo | Group 7: VX-661 100 mg qd | Total
Number analyzed (Participants) | 33 | 8 | 8 | 18 | 8 | 19 | 17 | 9 | 17 | 19 | 16 | 4 | 14 | 190
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8.42) | 35.3 (8.26) | 30.8 (6.63) | 28.3 (7.05) | 29.1 (7.12) | 29.2 (6.39) | 31 (9.3) | 28.2 (8.6) | 28.2 (6.46) | 27.9 (5.58) | 32.8 (11.92) | 34.5 (7.59) | 26.6 (7.01) | 29.8 (7.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 4 | 4 | 6 | 3 | 6 | 11 | 3 | 10 | 7 | 7 | 3 | 6 | 83
  Male | 20 | 4 | 4 | 12 | 5 | 13 | 6 | 6 | 7 | 12 | 9 | 1 | 8 | 107

OUTCOME MEASURES:

1. Primary Outcome: Safety as Determined by Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the Informed Consent Form is signed. AE includes serious as well as non-serious AEs. Serious Adverse Event (SAE) is any AE that results in any of the following: death; life-threatening condition; inpatient hospitalization or prolongation of hospitalization; persistent or significant disability or incapacity; congenital anomaly or birth defect; or other important medical event. Treatment-emergent adverse events are defined as adverse events that were reported or worsened on or after start of study drug through the Follow-up Visit (28 days after last dose of study drug) or premature discontinuation.
Time Frame: Start of study drug through the Follow-up Visit (Up to Day 56)
Population: Analysis was done using safety set which included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Group 1-6d Combined: Placebo | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 7: Placebo | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 33 | 8 | 8 | 18 | 8 | 19 | 17 | 9 | 17 | 19 | 16 | 4 | 14
participants
  Participants with AEs | 30 | 8 | 7 | 15 | 7 | 18 | 10 | 8 | 17 | 16 | 16 | 2 | 12
  Participants with SAEs | 5 | 1 | 1 | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 2 | 0 | 1

2. Primary Outcome: Change in Sweat Chloride From Baseline Through Study Day 28 for Group 1-5b
Description: Sweat samples were collected using an approved collection device. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug.
Time Frame: Baseline through Day 28
Population: The analysis was done using Full Analysis Set (FAS) which included all randomized participants who received at least 1 dose of study drug. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Groups:
- Group 1-5b Combined Placebo: All participants in group 1, 2a, 2b, 3a, 3b, 4, 5a and 5b who received placebo matched to VX-661 tablet and/or placebo matched to ivacaftor tablet for up to 28 days.
Arm/Group | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 1-5b Combined Placebo
Number analyzed (Participants) | 8 | 6 | 18 | 8 | 18 | 17 | 9 | 17 | 24
millimole per liter (mmol/L) | 3.92 [-0.5 to 8.34] | -4.76 [-9.75 to 0.22] | -5.06 [-8.02 to -2.09] | -20.43 [-24.75 to -16.12] | -6 [-8.98 to 3.02] | -6.04 [-9.12 to -2.96] | -10.46 [-14.53 to -6.39] | -2.63 [-5.67 to 0.41] | -0.86 [-3.36 to 1.65]
Statistical Analysis 1: Comparison: Group 1: VX-661 10 mg qd vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.0647, Mixed-effect repeated measure (MMRM); Least Squares (LS) Mean Difference = 4.77, 95% CI 2-sided [-0.3 to 9.84]
Statistical Analysis 2: Comparison: Group 2a: VX-661 30 mg qd vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.1686, MMRM; LS Mean Difference = -3.91, 95% CI 2-sided [-9.5 to 1.68]
Statistical Analysis 3: Comparison: Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.0348, MMRM; LS Mean Difference = -4.2, 95% CI 2-sided [-8.1 to -0.31]
Statistical Analysis 4: Comparison: Group 3a: VX-661 100 mg qd vs Group 1-5b Combined Placebo; Test type: Superiority; p < 0.0001, MMRM; LS Mean Difference = -19.58, 95% CI 2-sided [-24.57 to -14.59]
Statistical Analysis 5: Comparison: Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.0101, MMRM; LS Mean Difference = -5.14, 95% CI 2-sided [-9.03 to -1.25]
Statistical Analysis 6: Comparison: Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.011, MMRM; LS Mean Difference = -5.19, 95% CI 2-sided [-9.16 to -1.21]
Statistical Analysis 7: Comparison: Group 5a: VX-661 150 mg qd vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.0001, MMRM; LS Mean Difference = -9.6, 95% CI 2-sided [-14.38 to -4.82]
Statistical Analysis 8: Comparison: Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h vs Group 1-5b Combined Placebo; Test type: Superiority; p = 0.3745, MMRM; LS Mean Difference = -1.77, 95% CI 2-sided [-5.71 to 2.17]

3. Primary Outcome: Change in Sweat Chloride From Baseline Through Study Day 28 for Group 6
Description: Sweat samples were collected using an approved collection device. Baseline was defined as the most recent non-missing measurement collected before initial administration of study drug. As per planned analysis, participants who received placebo in Group 4 and 6 were combined and compared with Group 6.
Time Frame: Baseline through Day 28
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h: All participants in group 6d who received VX-661 50 mg tablet q12h and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
- Group 4 and 6 Combined: Placebo: All participants in group 4, 6a and 6d who received placebo matched to VX-661 tablet and/or placebo matched to ivacaftor tablet for up to 28 days.
Arm/Group | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 4 and 6 Combined: Placebo
Number analyzed (Participants) | 18 | 16 | 14
mmol/L | -6.07 [-10.84 to -1.31] | -7.89 [-12.3 to -3.48] | -1.19 [-5.5 to 3.12]
Statistical Analysis 1: Comparison: Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h vs Group 4 and 6 Combined: Placebo; Test type: Superiority; p = 0.0357, MMRM; LS Mean Difference = -6.7, 95% CI 2-sided [-12.94 to -0.46]

4. Primary Outcome: Change in Sweat Chloride From Baseline Through Study Day 28 for Group 7
Description: as for outcome 2
Time Frame: Baseline through Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Group 7: Placebo | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 4 | 13
mmol/L | 10.18 [-2.48 to 22.84] | -7.02 [-14.15 to 0.11]
Statistical Analysis 1: Comparison: Group 7: Placebo vs Group 7: VX-661 100 mg qd; Test type: Superiority; p = 0.0238, MMRM; LS Mean Difference = -17.2, 95% CI 2-sided [-31.75 to -2.65]

5. Secondary Outcome: Change in Sweat Chloride From Baseline to Each Visit up to Study Day 28 for Group 1-5b
Description: as for outcome 2
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each arm, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 1-5b Combined Placebo
Number analyzed (Participants) | 8 | 8 | 18 | 8 | 18 | 17 | 9 | 17 | 24
mmol/L
  Day 7: number analyzed (Participants) | 8 | 6 | 16 | 8 | 16 | 16 | 9 | 17 | 23
  Day 7 | 1.73 [-3.82 to 7.29] | -3.13 [-9.5 to 3.25] | -5.37 [-9.24 to -1.49] | -19.48 [-25 to -13.97] | -5.02 [-8.85 to -1.19] | -6.85 [-10.72 to -2.99] | -13.89 [-19.09 to -8.69] | -0.59 [-4.38 to 3.2] | 0.22 [-3.01 to 3.45]
  Day 14: number analyzed (Participants) | 8 | 6 | 17 | 8 | 14 | 14 | 9 | 15 | 24
  Day 14 | 0.91 [-4.64 to 6.46] | -7.88 [-14.25 to -1.5] | -6.55 [-10.34 to -2.76] | -28.23 [-33.75 to 22.72] | -6.77 [-10.81 to -2.74] | -7.37 [-11.44 to -3.3] | -10.28 [-15.48 to -5.08] | -2.4 [-6.38 to 1.58] | -1.32 [-4.5 to 1.87]
  Day 21: number analyzed (Participants) | 7 | 6 | 17 | 8 | 15 | 13 | 9 | 15 | 23
  Day 21 | 4.84 [-0.99 to 10.66] | -4.61 [-10.98 to 1.76] | -3.7 [-7.48 to 0.09] | -18.78 [-24.3 to -13.27] | -5.83 [-9.77 to -1.89] | -4.26 [-8.44 to -0.08] | -12.17 [-17.37 to -6.97] | -3.9 [-7.88 to 0.08] | -1.05 [-4.29 to 2.18]
  Day 28: number analyzed (Participants) | 7 | 6 | 17 | 8 | 16 | 14 | 9 | 15 | 22
  Day 28 | 8.19 [2.37 to 14.02] | -3.44 [-9.82 to 2.93] | -4.62 [-8.41 to -0.83] | -15.23 [-20.75 to -9.72] | -6.37 [-10.22 to -2.52] | -5.68 [-9.76 to -1.61] | -5.5 [-10.7 to 0.3] | -3.62 [-7.6 to 0.36] | -1.27 [-4.55 to 2.01]

6. Secondary Outcome: Change in Sweat Chloride From Baseline to Each Visit up to Study Day 28 for Group 6
Description: as for outcome 3
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug. Here, 'Number of participants analyzed' = those participants who were evaluable for this endpoint and 'Number Analyzed' = those participants who were evaluable at the specified time points for each group, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 4 and 6 Combined: Placebo
Number analyzed (Participants) | 19 | 16 | 14
mmol/L
  Day 7: number analyzed (Participants) | 15 | 13 | 13
  Day 7 | -6.61 [-12.06 to -1.16] | -11.04 [-16.37 to -5.7] | -0.36 [-5.54 to 4.83]
  Day 14: number analyzed (Participants) | 17 | 14 | 14
  Day 14 | -7.9 [-13.25 to -2.55] | -7.11 [-12.34 to -1.88] | -2.1 [-7.19 to 2.98]
  Day 21: number analyzed (Participants) | 13 | 14 | 13
  Day 21 | -6.34 [-12 to 0.68] | -6.98 [-12.2 to -1.76] | -2.47 [-7.67 to 2.72]
  Day 28: number analyzed (Participants) | 16 | 15 | 13
  Day 28 | -3.44 [-8.85 to 1.97] | -6.43 [-11.55 to -1.31] | 0.19 [-5.01 to 5.39]

7. Secondary Outcome: Change in Sweat Chloride From Baseline to Each Visit up to Study Day 28 for Group 7
Description: as for outcome 2
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug. Here, 'Number Analyzed' = those participants who were evaluable at the specified time points for each group, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Group 7: Placebo | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 4 | 14
mmol/L
  Day 7: number analyzed (Participants) | 4 | 12
  Day 7 | 4.87 [-8.32 to 18.06] | -7.28 [-14.76 to 0.2]
  Day 14: number analyzed (Participants) | 4 | 11
  Day 14 | 10.75 [-2.44 to 23.94] | -8.95 [-16.54 to -1.35]
  Day 21: number analyzed (Participants) | 4 | 10
  Day 21 | 9.37 [-3.82 to 22.56] | -4.14 [-11.86 to 3.58]
  Day 28: number analyzed (Participants) | 3 | 11
  Day 28 | 15.73 [1.85 to 29.61] | -7.72 [-15.31 to -0.13]

8. Secondary Outcome: Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 1-5b
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Arm/Group | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 1-5b Combined Placebo
Number analyzed (Participants) | 8 | 8 | 18 | 8 | 19 | 17 | 9 | 17 | 24
percent predicted of FEV1
  Post-Baseline Through Day 28 | 3.49 [0.21 to 6.77] | 1.63 [-1.62 to 4.87] | 1.3 [-0.87 to 3.47] | 1.6 [-1.64 to 4.85] | 2.9 [0.76 to 5.03] | 3.75 [1.47 to 6.02] | 2.54 [-0.53 to 5.61] | 3.61 [1.36 to 5.86] | -0.14 [-2.02 to 1.74]
  Day 7 | 2.72 [-1.17 to 6.62] | 0.8 [-3.09 to 4.69] | 0.47 [-2.13 to 3.06] | 3 [-0.89 to 6.89] | 2.9 [0.37 to 5.42] | 2.66 [-0.01 to 5.33] | 0.5 [-3.17 to 4.18] | 2.51 [-0.16 to 5.18] | -0.41 [-2.66 to 1.84]
  Day 14: number analyzed (Participants) | 8 | 8 | 18 | 8 | 18 | 15 | 8 | 16 | 24
  Day 14 | 5.25 [1.35 to 9.15] | 3.72 [-0.17 to 7.61] | 0.91 [-1.69 to 3.5] | 1.61 [-2.28 to 5.5] | 1.79 [-0.78 to 4.36] | 4.52 [1.73 to 7.3] | 2.79 [-1 to 6.59] | 3.72 [1 to 6.44] | 0.03 [-2.21 to 2.28]
  Day 21: number analyzed (Participants) | 7 | 8 | 18 | 8 | 17 | 15 | 9 | 16 | 24
  Day 21 | 2.71 [-1.34 to 6.76] | 1.8 [-2.09 to 5.69] | 1.84 [-0.75 to 4.44] | 0.25 [-3.64 to 4.15] | 3.88 [1.27 to 6.5] | 3.37 [0.58 to 6.15] | 4.52 [0.85 to 8.19] | 4.08 [1.36 to 6.8] | 0.18 [-2.07 to 2.43]
  Day 28: number analyzed (Participants) | 7 | 8 | 17 | 8 | 17 | 15 | 9 | 16 | 23
  Day 28 | 3.26 [-0.79 to 7.32] | 0.19 [-3.7 to 4.08] | 1.99 [-0.65 to 4.63] | 1.55 [-2.34 to 5.45] | 3.02 [0.4 to 5.63] | 4.44 [1.66 to 7.23] | 2.34 [-1.33 to 6.01] | 4.13 [1.41 to 6.86] | -0.36 [-2.63 to 1.92]

9. Secondary Outcome: Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 6
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. As per planned analysis, participants who received placebo in Group 4 and 6 were combined and compared with Group 6.
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Arm/Group | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 4 and 6 Combined: Placebo
Number analyzed (Participants) | 19 | 16 | 14
percent predicted of FEV1
  Post-Baseline Through Day 28: number analyzed (Participants) | 18 | 16 | 14
  Post-Baseline Through Day 28 | 0.94 [-1.42 to 3.3] | 2.31 [-0.19 to 4.8] | 1.47 [-1.2 to 4.13]
  Day 7: number analyzed (Participants) | 18 | 16 | 14
  Day 7 | 1.37 [-1.33 to 4.08] | 1.95 [-0.93 to 4.82] | 1.09 [-1.97 to 4.15]
  Day 14: number analyzed (Participants) | 17 | 16 | 14
  Day 14 | 1.2 [-1.55 to 3.95] | 2.52 [-0.36 to 5.4] | 1.37 [-1.69 to 4.44]
  Day 21: number analyzed (Participants) | 17 | 16 | 13
  Day 21 | 0.36 [-2.38 to 3.11] | 3.21 [0.33 to 6.08] | 1.73 [-1.39 to 4.85]
  Day 28: number analyzed (Participants) | 16 | 16 | 13
  Day 28 | 0.81 [-1.97 to 3.6] | 1.56 [-1.32 to 4.44] | 1.67 [-1.45 to 4.8]

10. Secondary Outcome: Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 7
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted of FEV1
Arm/Group | Group 7: Placebo | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 4 | 14
percent predicted of FEV1
  Post-Baseline Through Day 28 | 1.4 [-5.04 to 7.83] | 4.6 [1.17 to 8.03]
  Day 7 | 3 [-3.55 to 9.55] | 4.14 [0.65 to 7.63]
  Day 14 | 0.98 [-5.56 to 7.53] | 5.22 [1.73 to 8.71]
  Day 21 | 2.72 [-3.83 to 9.27] | 3.88 [0.39 to 7.38]
  Day 28 | -1.12 [-7.66 to 5.43] | 5.16 [1.67 to 8.65]

11. Secondary Outcome: Change in FEV1 (Liter [L]) From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 1-5b
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug. Here 'Number Analyzed' = those participants who were evaluable at the specified time points for each group, respectively.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 1-5b Combined Placebo
Number analyzed (Participants) | 8 | 8 | 18 | 8 | 19 | 17 | 9 | 17 | 24
Liters
  PB Through Day 28 | 0.14 [0.02 to 0.26] | 0.07 [-0.05 to 0.19] | 0.05 [-0.03 to 0.13] | 0.04 [-0.08 to 0.16] | 0.1 [0.02 to 0.18] | 0.14 [0.06 to 0.23] | 0.1 [-0.01 to 0.21] | 0.12 [0.04 to 0.21] | 0.01 [-0.06 to 0.08]
  Day 7 | 0.11 [-0.04 to 0.25] | 0.02 [-0.13 to 0.16] | 0.02 [-0.08 to 0.12] | 0.09 [-0.06 to 0.24] | 0.1 [0 to 0.19] | 0.11 [0.01 to 0.21] | 0.02 [-0.12 to 0.16] | 0.08 [-0.02 to 0.18] | -0.01 [-0.09 to 0.08]
  Day 14: number analyzed (Participants) | 8 | 8 | 18 | 8 | 18 | 15 | 8 | 16 | 24
  Day 14 | 0.2 [0.05 to 0.34] | 0.14 [-0.01 to 0.28] | 0.03 [-0.07 to 0.12] | 0.04 [-0.11 to 0.19] | 0.05 [-0.04 to 0.15] | 0.17 [0.06 to 0.27] | 0.11 [-0.03 to 0.25] | 0.12 [0.02 to 0.23] | 0.02 [-0.07 to 0.1]
  Day 21: number analyzed (Participants) | 7 | 8 | 18 | 8 | 17 | 15 | 9 | 16 | 24
  Day 21 | 0.12 [-0.03 to 0.27] | 0.08 [-0.06 to 0.23] | 0.07 [-0.03 to 0.17] | 0 [-0.15 to 0.15] | 0.14 [0.04 to 0.23] | 0.13 [0.02 to 0.23] | 0.18 [0.04 to 0.31] | 0.14 [0.04 to 0.24] | 0.02 [-0.06 to 0.1]
  Day 28: number analyzed (Participants) | 7 | 8 | 17 | 8 | 17 | 15 | 9 | 16 | 23
  Day 28 | 0.13 [-0.02 to 0.28] | 0.03 [-0.11 to 0.18] | 0.08 [-0.02 to 0.18] | 0.04 [-0.11 to 0.18] | 0.1 [0.01 to 0.2] | 0.16 [0.06 to 0.27] | 0.09 [-0.05 to 0.23] | 0.15 [0.05 to 0.26] | 0.01 [-0.08 to 0.09]

12. Secondary Outcome: Change in FEV1 (L) From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 6
Description: as for outcome 9
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 4 and 6 Combined: Placebo
Number analyzed (Participants) | 19 | 16 | 14
Liters
  Post-Baseline Through Day 28: number analyzed (Participants) | 18 | 16 | 14
  Post-Baseline Through Day 28 | 0.02 [-0.07 to 0.11] | 0.09 [-0.01 to 0.18] | 0.07 [-0.04 to 0.17]
  Day 7: number analyzed (Participants) | 18 | 16 | 14
  Day 7 | 0.04 [-0.07 to 0.14] | 0.06 [-0.05 to 0.17] | 0.05 [-0.06 to 0.17]
  Day 14: number analyzed (Participants) | 17 | 16 | 14
  Day 14 | 0.03 [-0.07 to 0.14] | 0.1 [-0.01 to 0.21] | 0.06 [-0.05 to 0.18]
  Day 21: number analyzed (Participants) | 17 | 16 | 13
  Day 21 | -0.01 [-0.11 to 0.1] | 0.13 [0.02 to 0.24] | 0.08 [-0.04 to 0.2]
  Day 28: number analyzed (Participants) | 16 | 16 | 13
  Day 28 | 0.02 [-0.08 to 0.13] | 0.06 [-0.05 to 0.17] | 0.08 [-0.04 to 0.2]

13. Secondary Outcome: Change in FEV1 (L) From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 7
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: Baseline, Day 7, Day 14, Day 21, Day 28
Population: The analysis was done using FAS which included all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Group 7: Placebo | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 4 | 14
Liters
  Post-Baseline Through Day 28 | 0.09 [-0.16 to 0.34] | 0.16 [0.03 to 0.29]
  Day 7 | 0.14 [-0.11 to 0.39] | 0.15 [0.01 to 0.28]
  Day 14 | 0.08 [-0.17 to 0.33] | 0.18 [0.05 to 0.32]
  Day 21 | 0.14 [-0.11 to 0.4] | 0.13 [-0.01 to 0.26]
  Day 28 | -0.01 [-0.26 to 0.25] | 0.19 [0.05 to 0.32]

14. Secondary Outcome: Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 1-5b
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: Baseline, Day 14, Day 28
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 1-5b Combined Placebo
Number analyzed (Participants) | 8 | 8 | 18 | 8 | 19 | 17 | 9 | 17 | 24
units on a scale
  PB Through Day 28: number analyzed (Participants) | 8 | 8 | 18 | 8 | 18 | 15 | 9 | 16 | 24
  PB Through Day 28 | 4.02 [-4.38 to 12.43] | 5.54 [-2.72 to 13.79] | 3.8 [-1.74 to 9.35] | 0.61 [-7.64 to 8.86] | 3.52 [-2.02 to 9.06] | 5.15 [-0.88 to 11.19] | 2.58 [-5.21 to 10.37] | 7.62 [1.78 to 13.45] | 1.69 [-3.1 to 6.48]
  Day 14: number analyzed (Participants) | 8 | 8 | 18 | 8 | 18 | 15 | 9 | 16 | 24
  Day 14 | 6.67 [-2.9 to 16.25] | 4.84 [-4.73 to 14.41] | 4.29 [-2.09 to 10.67] | 0.27 [-9.3 to 9.83] | 2.81 [-3.56 to 9.19] | 4.41 [-2.58 to 11.4] | 4.13 [-4.9 to 13.16] | 7.13 [0.37 to 13.89] | 0.53 [-4.99 to 6.05]
  Day 28: number analyzed (Participants) | 7 | 8 | 17 | 8 | 17 | 15 | 9 | 16 | 23
  Day 28 | 1.38 [-8.7 to 11.45] | 6.23 [-3.34 to 15.8] | 3.31 [-3.21 to 9.84] | 0.95 [-8.61 to 10.52] | 4.22 [-2.29 to 10.74] | 5.9 [-1.1 to 12.89] | 1.03 [-8 to 10.06] | 8.1 [1.34 to 14.87] | 2.85 [-2.76 to 8.46]

15. Secondary Outcome: Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 6
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms (for example, coughing, congestion, wheezing), score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life. As per planned analysis, participants who received placebo in Group 4 and 6 were combined and compared with Group 6.
Time Frame: Baseline, Day 14, Day 28
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 4 and 6 Combined: Placebo
Number analyzed (Participants) | 19 | 16 | 14
units on a scale
  Post-Baseline Through Day 28: number analyzed (Participants) | 17 | 16 | 14
  Post-Baseline Through Day 28 | 0.87 [-4.44 to 6.19] | 1.91 [-3.5 to 7.33] | 1.65 [-4.18 to 7.49]
  Day 14: number analyzed (Participants) | 17 | 16 | 14
  Day 14 | 2.02 [-3.97 to 8.02] | 0.87 [-5.25 to 6.99] | 2.78 [-3.76 to 9.32]
  Day 28: number analyzed (Participants) | 17 | 16 | 13
  Day 28 | -0.27 [-6.27 to 5.72] | 2.96 [-3.16 to 9.08] | 0.53 [-6.18 to 7.23]

16. Secondary Outcome: Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain Score From Baseline to Each Visit and From Baseline Through Study Day 28 for Group 7
Description: as for outcome 14
Time Frame: Baseline, Day 14, Day 28
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Group 7: Placebo | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 4 | 14
units on a scale
  Post-Baseline Through Day 28 | -3.02 [-13.52 to 7.47] | 3.79 [-1.78 to 9.36]
  Day 14: number analyzed (Participants) | 4 | 13
  Day 14 | 1.83 [-10.64 to 14.3] | 5.24 [-1.56 to 12.04]
  Day 28 | -7.87 [-20.34 to 4.6] | 2.33 [-4.24 to 8.91]

17. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to 24 Hours (AUC0-24h) of VX-661 After Administration of VX-661 Monotherapy
Description: Participants who received VX-661 monotherapy (Group 1, 2a, 3a and 5a) were analyzed for this outcome measure. PK analysis (AUC0-24h) was not planned for placebo reporting arms.
Time Frame: Day 28
Population: The analysis was done using Pharmacokinetics (PK) Set.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 3a: VX-661 100 mg qd | Group 5a: VX-661 150 mg qd
Number analyzed (Participants) | 7 | 8 | 8 | 9
nanogram*hour per milliliter (ng*hr/mL) | 6260 (2650) | 23000 (6550) | 88100 (51100) | 98900 (20200)

18. Secondary Outcome: AUC0-24h of VX-661 and AUC0-12h of Ivacaftor After Administration of VX-661 in Combination With Ivacaftor
Description: Participants who received VX-661 in combination with Ivacaftor (Group 2b, 3b, 4, 5b, 6a, 6d and 7) were analyzed for this outcome measure. PK analysis was not planned for placebo reporting arms.
Time Frame: Day 28
Population: The analysis was done using PK Set.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Groups:
- Group 5b: VX-661 150 mg qd/ Ivacaftor 150 mg q12h: All participants in group 5b who received VX-661 150 mg tablet qd and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
- Group 6a: VX-661 100 mg qd/ Ivacaftor 50 mg q12h: All participants in group 6a who received VX-661 100 mg tablet qd and Ivacaftor 50 mg tablet q12h orally for up to 28 days.
- Group 6d: VX-661 50 mg q12h/ Ivacaftor 150 mg q12h: All participants in group 6d who received VX-661 50 mg tablet and Ivacaftor 150 mg tablet q12h orally for up to 28 days.
- Group 7: VX-661 100 mg qd: All participants in group 7 who received VX-661 100 mg tablet orally qd in combination with physician prescribed Kalydeco for up to 28 days.
Arm/Group | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5b: VX-661 150 mg qd/ Ivacaftor 150 mg q12h | Group 6a: VX-661 100 mg qd/ Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/ Ivacaftor 150 mg q12h | Group 7: VX-661 100 mg qd
Number analyzed (Participants) | 17 | 13 | 15 | 16 | 17 | 15 | 14
ng*h/mL
  AUC0-24h of VX-661 | 8950 (2370) | 26300 (5870) | 82700 (23300) | 138000 (49700) | 77600 (17800) | 73300 (22900) | 90600 (30800)
  AUC0-12h of Ivacaftor: number analyzed (Participants) | 16 | 11 | 13 | 13 | 15 | 14 | 14
  AUC0-12h of Ivacaftor | 10100 (4380) | 11700 (4870) | 10900 (3890) | 16000 (10400) | 3690 (1460) | 11700 (5450) | 12400 (6170)

ADVERSE EVENTS:
Time Frame: Start of study drug through the Follow-up Visit (Up to Day 56)
Groups:
- Group 1: VX-661 10 mg qd: All participants in group 1 who received VX-661 10 milligram (mg) tablet orally qd for up to 28 days.
Arm/Group | Group 1-6d Combined: Placebo | Group 1: VX-661 10 mg qd | Group 2a: VX-661 30 mg qd | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h | Group 3a: VX-661 100 mg qd | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h | Group 5a: VX-661 150 mg qd | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h | Group 7: Placebo | Group 7: VX-661 100 mg qd
Serious Adverse Events (participants affected / at risk) | 5/33 | 1/8 | 1/8 | 1/18 | 0/8 | 2/19 | 2/17 | 0/9 | 0/17 | 1/19 | 2/16 | 0/4 | 1/14
Other Adverse Events (participants affected / at risk) | 30/33 | 8/8 | 7/8 | 15/18 | 7/8 | 18/19 | 9/17 | 8/9 | 17/17 | 16/19 | 16/16 | 2/4 | 12/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1-6d Combined: Placebo (N=33) | Group 1: VX-661 10 mg qd (N=8) | Group 2a: VX-661 30 mg qd (N=8) | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h (N=18) | Group 3a: VX-661 100 mg qd (N=8) | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h (N=19) | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h (N=17) | Group 5a: VX-661 150 mg qd (N=9) | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h (N=17) | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h (N=19) | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h (N=16) | Group 7: Placebo (N=4) | Group 7: VX-661 100 mg qd (N=14)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 5 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1-6d Combined: Placebo (N=33) | Group 1: VX-661 10 mg qd (N=8) | Group 2a: VX-661 30 mg qd (N=8) | Group 2b: VX-661 10 mg qd/Ivacaftor 150 mg q12h (N=18) | Group 3a: VX-661 100 mg qd (N=8) | Group 3b: VX-661 30 mg qd/Ivacaftor 150 mg q12h (N=19) | Group 4: VX-661 100 mg qd/Ivacaftor 150 mg q12h (N=17) | Group 5a: VX-661 150 mg qd (N=9) | Group 5b: VX-661 150 mg qd/Ivacaftor 150 mg q12h (N=17) | Group 6a: VX-661 100 mg qd/Ivacaftor 50 mg q12h (N=19) | Group 6d: VX-661 50 mg q12h/Ivacaftor 150 mg q12h (N=16) | Group 7: Placebo (N=4) | Group 7: VX-661 100 mg qd (N=14)
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 4 | 1 | 1 | 1 | 3 | 0 | 1 | 2 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 2
Application site rash (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site swelling (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Medical device complication (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thinking abnormal (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast tenderness (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Menstrual disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary function test decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal examination abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary casts present (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine colour abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3 | 2 | 2 | 3 | 2 | 2 | 3 | 4 | 3 | 0 | 4
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 2 | 1 | 2 | 3 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 8 | 1 | 1 | 2 | 1 | 4 | 0 | 1 | 2 | 4 | 4 | 0 | 3
Sinus headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 1 | 2 | 1 | 4 | 0 | 1 | 5 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin E deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin K deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 8 | 0 | 0 | 4 | 1 | 4 | 3 | 1 | 2 | 2 | 3 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 2 | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 3 | 1 | 1
Sinusitis (Infections and infestations) | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Pharmacokinetic (PK) final data are not yet available. Once the data are available for PK endpoints, the posting will be updated to include the same.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Restriction Description: PI is free to publish results of the study after (1)first multi-center publication, (2)if sponsor elects not to publish the results, or(3)18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.